CLINICAL TRIAL: NCT03877484
Title: A Prospective, Multi-center, Post-Market Clinical Follow-Up Study to Evaluate the Safety and Effectiveness of ALLEVYN Gentle Border
Brief Title: Evaluation of the Safety and Effectiveness of ALLEVYN Gentle Border
Status: Completed | Type: Observational
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Other Study IDs: ALLEV.PMCF.2017.13
Record Dates: First submitted 2019-02-06; First posted 2019-03-15 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2021-12

CONDITIONS: Wound
Keywords: chronic and acute wounds; full-thickness; partial thickness; shadow granulating; exuding wounds; including pressure ulcers; leg ulcers; diabetic foot ulcers; dehisced surgical wounds
MeSH Terms: conditions — Wounds and Injuries; Bronchiolitis Obliterans Syndrome; Leg Ulcer; Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ALLEVYN Gentle border — ALLEVYN Gentle border is a triple layer foam dressing consisting of a highly absorbent hydrocellular foam pad held between a perforated wound contact layer (WCL), which is coated with a soft silicone gel adhesive and a highly permeable outer top film.

SUMMARY:
The clinical study will evaluate the safety and effectiveness of the ALLEVYN Gentle Border. The study is a post-market clinical follow-up to assess clinical performance and safety of ALLEVYN Gentle Border with new wound contact layer to support performance claims.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. 18 years of age or older.
3. Willing and able to make all required study visits.
4. Able to follow instructions and deemed capable of completing the CWIS questionnaire, Patient Assessment Scale and Pain Scale.
5. Presence of a moderately to highly exuding wound of at least 3cm2 in size.
6. Presence of a chronic wound of at least 6 weeks duration at the point of enrollment; full-thickness, partial thickness or shallow granulating wounds.

   Chronic wounds include:
   * pressure ulcers or
   * leg ulcers or
   * diabetic foot ulcers

   or

   Presence of an acute wound at the point of enrollment; full thickness, partial thickness or shallow granulating wounds

   Acute wounds include:
   * dehisced surgical or
   * traumatic wounds
7. The patient has a wound size which can be treated with the available sizes and shapes of ALLEVYN Gentle Border. Cutting of the dressing is allowed, if needed. ALLEVYN Gentle Border can be cut and an aseptic technique should be used with cutting the dressing. Ensure any exposed foam areas are covered with an appropriate film dressing taking care not to cover the entire dressing.

Exclusion Criteria:

1. Subjects with confirmed or suspected clinically infected reference wound.
2. Reference wound undergoing treatment with compression therapy.
3. Contraindications or hypersensitivity to the use of the ALLEVYN Gentle Border.
4. Participation in the treatment period of another clinical trial within 30 days of Visit 1 or planned participation overlapping with this study.
5. Subjects with skin features (e.g. tattoos, skin color, pre-existing scarring) which, in the opinion of the Investigator, could interfere with the study assessments.
6. Subjects who have participated previously in this clinical trial.
7. Subjects with a history of poor compliance with medical treatment.
8. Subjects with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Forty adult subjects with moderate to highly exuding wounds that require a dressing will be recruited. Only subjects with acute wounds or chronic wounds which are present > 6 weeks will be enrolled. Chronic wounds will include pressure ulcers, leg ulcers, diabetic foot ulcers. Acute wounds will include dehisced surgical or traumatic wounds. In order to ensure a balanced distribution on chronic and acute indications, at least 10 subjects with chronic wounds and at least 10 subjects with acute wounds will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Reinhold, MD, Principal Investigator — VZ Dermatologisches Zentrum Bonn; Cornelia Erfurt-Berge, MD, Principal Investigator — University Hospital Erlangen, Department of Dermatology; Ulrike Raap, MD, Principal Investigator — Klinikum Oldenburg, Universitätsklinik für Dermatologie und Allergologie
Locations (6):
- Centre Hospitalier William Morey, Chalon-sur-Saône, France
- Germany (4):
  - MVZ Dermatologisches Zentrum Bonn GmbH, Bonn
  - University Hospital Erlangen, Department of Dermatology, Erlangen
  - Niels-Stensen-Kliniken Christliches Klinikum Melle GmbH, Melle
  - Klinikum Oldenburg, University Clinic for Dermatology and Allergy, Oldenburg
- Northumbria Healthcare NHS Foundation Trust, Ashington, Northumberland, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants were terminated prior to study treatment, following consent, and did not meet eligibility criteria.
Period: Overall Study
Arm/Group | ALLEVYN Gentle Border
Started | 40
Completed | 30
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (18.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 38
  Race/Ethnicity: Missing | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.1 (6.1)
Wound Type [Count of Participants; unit: Participants]
  Acute | 14
  Chronic | 26
Wound Duration [Mean (Standard Deviation); unit: days] | 158.3 (266.4)
Wound Area [Mean (Standard Deviation); unit: cm^2] | 11.9 (13.8)
Exudate Levels [Count of Participants; unit: Participants]
  None | 6
  Scant | 4
  Small | 17
  Moderate | 11
  Large | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Wound Area From Baseline to End of Study Visit
Description: Change in wound area from baseline to end of study visit at 28 days was measured by wound photographs from a specific digital camera that standardized and calculated wound length, width, and depth automatically.
Time Frame: Baseline through 28 days (±3 days).
Population: All participants enrolled in the study that completed at least one post-baseline assessment for the specified outcome with available data at the time frame indicated using the last observation carried forward (LOCF).
Measure: Median (95% Confidence Interval); unit: square centimeters (cm^2)
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 40
square centimeters (cm^2) | 2.2 [0.9 to 3.9]

2. Secondary Outcome: Change in Wound Area From Baseline to 7 Days (±3 Days), 14 Days (±3 Days), and 21 Days (±3 Days)
Description: Change in wound area from baseline to 7 days, 14 days and 21 days. Wound area was measured by photographs from a specific digital camera that standardized and calculated wound length, width, and depth automatically.
Time Frame: Baseline to 7 days (±3 days), 14 days (±3 days), and 21 days (±3 days)
Population: All participants enrolled in the study that completed at least one post-baseline assessment for the specified outcome with available data at the time frame indicated.
Measure: Median (95% Confidence Interval); unit: square centimeters (cm^2)
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 37
square centimeters (cm^2)
  Baseline to 7 days (±3 days) | 0.5 [-0.2 to 0.8]
  Baseline to 14 days (±3 days): number analyzed (Participants) | 34
  Baseline to 14 days (±3 days) | 1.2 [0.5 to 2.1]
  Baseline to 21 days (±3 days): number analyzed (Participants) | 32
  Baseline to 21 days (±3 days) | 1.7 [0.6 to 3.1]

3. Secondary Outcome: Change in Wound Depth From Baseline to 7 Days (±3 Days), 14 Days (±3 Days), 21 Days (±3 Days) and 28 Days (±3 Days)
Description: Wound depth at baseline, 7, 14, 21 and 28 days were measured by wound photographs from a specific digital camera that standardized and calculated wound length, width, and depth automatically.
Time Frame: Baseline, 7 days, 14 days, 21 days, 28 days
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: millimeters (mm)
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 34
millimeters (mm)
  Baseline to 7 Days | 0.1 [0.01 to 0.3]
  Baseline to 14 Days: number analyzed (Participants) | 29
  Baseline to 14 Days | 0.1 [-0.01 to 0.3]
  Baseline to 21 Days: number analyzed (Participants) | 25
  Baseline to 21 Days | 0.1 [-0.01 to 0.6]
  Baseline to 28 Days: number analyzed (Participants) | 22
  Baseline to 28 Days | 0.1 [-0.01 to 0.6]

4. Secondary Outcome: Change in Wound Volume From Baseline to 7 Days (±3 Days), 14 Days (±3 Days), 21 Days (±3 Days) and 28 Days (±3 Days)
Description: Change in exudate wound volume measured from baseline to 7 days, 14 days, 21 days and 28 days.
Time Frame: Baseline, 7 days, 14 days, 21 days, and 28 days
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: cubic centimeter (cm^3)
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 34
cubic centimeter (cm^3)
  Baseline to 7 Days (±3 Days) | 0.07 [-0.01 to 0.2]
  Baseline to 14 Days (±3 Days): number analyzed (Participants) | 29
  Baseline to 14 Days (±3 Days) | 0.08 [-0.01 to 0.2]
  Baseline to 21 Days (±3 Days): number analyzed (Participants) | 25
  Baseline to 21 Days (±3 Days) | 0.1 [0.01 to 0.3]
  Baseline to 28 Days (±3 Days): number analyzed (Participants) | 22
  Baseline to 28 Days (±3 Days) | 0.1 [0.02 to 0.3]

5. Secondary Outcome: Percentage Change in Wound Area From Baseline to 7 Days (±3 Days), 14 Days (±3 Days), and 21 Days (±3 Days)
Description: Percentage change in wound area from baseline visit to visits 2 (7 Days), 3 (14 days) and 4 (21 days).
Time Frame: Baseline to 7 days (±3 days), 14 days (±3 days), and 21 days (±3 days)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: percent change in wound area
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 37
percent change in wound area
  Baseline to 7 days (±3 days) | 9.5 [-37.9 to 91.8]
  Baseline to 14 days (±3 days): number analyzed (Participants) | 34
  Baseline to 14 days (±3 days) | 21.3 [-118.8 to 100]
  Baseline to 21 days (±3 days): number analyzed (Participants) | 32
  Baseline to 21 days (±3 days) | 40.8 [-152.8 to 100]
  Baseline to 28 Days: number analyzed (Participants) | 30
  Baseline to 28 Days | 49.9 [-114 to 100]

6. Secondary Outcome: Percentage Change in Wound Depth From Baseline to 7 Days (±3 Days), 14 Days (±3 Days), and 21 Days (±3 Days)
Description: Percentage change in wound depth from baseline visit to visits 2 (7 Days), 3 (14 days) and 4 (21 days).
Time Frame: Baseline to 7 days (±3 days), 14 days (±3 days), and 21 days (±3 days)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: percent change in wound depth
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 34
percent change in wound depth
  Baseline to 7 days (±3 days) | 29.1 [-4402.2 to 94.6]
  Baseline to 14 days (±3 days): number analyzed (Participants) | 29
  Baseline to 14 days (±3 days) | 34.7 [-1306 to 100]
  Baseline to 21 days (±3 days): number analyzed (Participants) | 25
  Baseline to 21 days (±3 days) | 40 [-3795.5 to 100]
  Baseline to 28 Days (±3 days): number analyzed (Participants) | 22
  Baseline to 28 Days (±3 days) | 27.7 [-1433.9 to 100]

7. Secondary Outcome: Percentage Change in Wound Volume From Baseline to 7 Days (±3 Days), 14 Days (±3 Days), and 21 Days (±3 Days)
Description: Percentage change in wound volume from baseline visit to visits 2 (7 Days), 3 (14 days) and 4 (21 days).
Time Frame: Baseline to 7 days (±3 days), 14 days (±3 days), and 21 days (±3 days)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: percent change in wound volume
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 34
percent change in wound volume
  Baseline to 7 days (±3 days) | 38.7 [-5023.5 to 97.6]
  Baseline to 14 days (±3 days): number analyzed (Participants) | 29
  Baseline to 14 days (±3 days) | 21.3 [-118.8 to 100]
  Baseline to 21 days (±3 days): number analyzed (Participants) | 25
  Baseline to 21 days (±3 days) | 40.8 [-152.8 to 100]
  Baseline to 28 Days (±3 days): number analyzed (Participants) | 22
  Baseline to 28 Days (±3 days) | 49.9 [-114 to 100]

8. Secondary Outcome: Exudate Management: Number of Dressings With Leakage
Description: The count of dressings applied on participants with exudate present that experienced any dressing leakage (Yes/No).
Time Frame: Dressing application to removal, up to 7 days (±3 Days)
Population: Only participants enrolled in the study with any Exudate Levels present (i.e., scant, small, moderate, or large) that completed at least one post-baseline assessment for the specified outcome with available data at the time frame indicated. Of the 40 participants enrolled, 34 participants had exudate present.
Measure: Count of Units; unit: dressings
Units Other Than Participants: dressings
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 34
Number analyzed (dressings) | 242
dressings
  Any Dressing Leakage: Yes | 34
  Any Dressing Leakage: No | 208

9. Secondary Outcome: Exudate Amount at 7 Days (±3 Days), 14 Days (±3 Days), 21 Days (±3 Days) and 28 Days (±3 Days)
Description: Count of participants with wound exudate amounts identified as:
  * None
  * Scant
  * Small
  * Moderate
  * Large
Time Frame: 7 days (±3 Days), 14 days (±3 Days), 21 days (±3 Days), and 28 days (±3 Days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 40
Participants
  7 days (±3 Days): None | 5
  7 days (±3 Days): Scant | 4
  7 days (±3 Days): Small | 13
  7 days (±3 Days): Moderate | 16
  7 days (±3 Days): Large | 2
  14 days (±3 Days): None | 7
  14 days (±3 Days): Scant | 2
  14 days (±3 Days): Small | 19
  14 days (±3 Days): Moderate | 11
  14 days (±3 Days): Large | 1
  21 days (±3 Days): None | 7
  21 days (±3 Days): Scant | 2
  21 days (±3 Days): Small | 20
  21 days (±3 Days): Moderate | 9
  21 days (±3 Days): Large | 2
  28 days (±3 Days): None | 8
  28 days (±3 Days): Scant | 3
  28 days (±3 Days): Small | 17
  28 days (±3 Days): Moderate | 8
  28 days (±3 Days): Large | 4

10. Secondary Outcome: Exudate Type at 7 (±3 Days), 14 (±3 Days), 21 (±3 Days) and 28 Days (±3 Days)
Description: Count of participants with wound exudate types identified as:
  * None
  * Bloody
  * Serosanguineous
  * Serous
  * Purulent
Time Frame: 7 days (±3 Days), 14 days (±3 Days), 21 days (±3 Days), and 28 days (±3 Days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 40
Participants
  7 days (±3 Days): None | 5
  7 days (±3 Days): Bloody | 1
  7 days (±3 Days): Serosanguineous | 20
  7 days (±3 Days): Serous | 11
  7 days (±3 Days): Purulent | 3
  14 days (±3 Days): None | 7
  14 days (±3 Days): Bloody | 1
  14 days (±3 Days): Serosanguineous | 19
  14 days (±3 Days): Serous | 7
  14 days (±3 Days): Purulent | 6
  21 days (±3 Days): None | 7
  21 days (±3 Days): Bloody | 1
  21 days (±3 Days): Serosanguineous | 21
  21 days (±3 Days): Serous | 7
  21 days (±3 Days): Purulent | 4
  28 days (±3 Days): None | 8
  28 days (±3 Days): Bloody | 0
  28 days (±3 Days): Serosanguineous | 19
  28 days (±3 Days): Serous | 9
  28 days (±3 Days): Purulent | 4

11. Secondary Outcome: Level of Wound Odour at Baseline, 7 Days (±3 Days), 14 Days (±3 Days), 21 Days (±3 Days) and 28 Days (±3 Days)
Description: Count of participants level of odour at baseline, 7 Days (±3 Days), 14 Days (±3 Days), 21 Days (±3 Days), and 28 Days (±3 Days) identified as:
  * None
  * Mild
  * Moderate
  * Strong
Time Frame: Baseline, 7 days (±3 Days), 14 days (±3 Days), 21 days (±3 Days), 28 days (±3 Days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 40
Participants
  Baseline: None | 34
  Baseline: Mild | 5
  Baseline: Moderate | 0
  Baseline: Strong | 1
  7 days (±3 Days): None | 34
  7 days (±3 Days): Mild | 6
  7 days (±3 Days): Moderate | 0
  7 days (±3 Days): Strong | 0
  14 days (±3 Days): number analyzed (Participants) | 36
  14 days (±3 Days): None | 30
  14 days (±3 Days): Mild | 6
  14 days (±3 Days): Moderate | 0
  14 days (±3 Days): Strong | 0
  21 days (±3 Days): number analyzed (Participants) | 32
  21 days (±3 Days): None | 26
  21 days (±3 Days): Mild | 6
  21 days (±3 Days): Moderate | 0
  21 days (±3 Days): Strong | 0
  28 days (±3 Days): number analyzed (Participants) | 30
  28 days (±3 Days): None | 26
  28 days (±3 Days): Mild | 4
  28 days (±3 Days): Moderate | 0
  28 days (±3 Days): Strong | 0

12. Secondary Outcome: Reason for Dressing Change
Description: Overall frequency of dressing changes categorized with the following reasons(Yes/No):
  * Reason for dressing change routine
  * ALLEVYN been in place 7 days
  * Dressing saturated
  * Strikethrough
  * Leakage
  * Pain
  * Dressing fell off
  * Dressing got wet during shower/bathing
  * Subject removed dressing
  * Other
Time Frame: Upon dressing removal, up to 7 days (±3 Days)
Population: as for outcome 2
Measure: Count of Units; unit: dressings
Units Other Than Participants: dressings
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 39
Number analyzed (dressings) | 222
dressings
  Reason for dressing change routine: number analyzed (dressings) | 106
  Reason for dressing change routine: No | 34
  Reason for dressing change routine: Yes | 72
  ALLEVYN been in place 7 days: No | 195
  ALLEVYN been in place 7 days: Yes | 27
  Dressing saturated: No | 195
  Dressing saturated: Yes | 27
  Strikethrough: No | 197
  Strikethrough: Yes | 25
  Leakage: No | 212
  Leakage: Yes | 10
  Pain: No | 221
  Pain: Yes | 1
  Dressing fell off: No | 215
  Dressing fell off: Yes | 7
  Dressing got wet during shower/bathing: No | 220
  Dressing got wet during shower/bathing: Yes | 2
  Subject removed dressing: No | 221
  Subject removed dressing: Yes | 1
  Other: No | 146
  Other: Yes | 76

13. Secondary Outcome: Condition of Surrounding Skin
Description: The condition of surrounding skin (i.e., peri-wound) was assessed to ensure there was no compromise to skin condition as a result of dressing wear, which could impact the wound healing progress. Number of participants condition of the peri-wound was classified as:
  * Normal
  * Erythematous
  * 50% to <75% wound covered
  * 25% to <50% wound covered
  * <25% wound covered
  * Missing
Time Frame: Baseline and 28 days (±3 Days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 40
Participants
  Baseline: Normal | 22
  Baseline: Erythematous | 14
  Baseline: 50% to <75% wound covered | 0
  Baseline: 25% to <50% wound covered | 0
  Baseline: <25% wound covered | 4
  Baseline: Missing | 0
  28 days (±3 Days): number analyzed (Participants) | 30
  28 days (±3 Days): Normal | 18
  28 days (±3 Days): Erythematous | 9
  28 days (±3 Days): 50% to <75% wound covered | 1
  28 days (±3 Days): 25% to <50% wound covered | 0
  28 days (±3 Days): <25% wound covered | 0
  28 days (±3 Days): Missing | 2

14. Secondary Outcome: Signs of Clinical Infection
Description: Any signs of clinical infection (Yes/No) identified at 7 Days (±3 Days), 14 Days (±3 Days), 21 Days (±3 Days) and 28 Day (±3 Days) visits.
Time Frame: 7 days (±3 Days), 14 days (±3 Days), 21 days (±3 Days), 28 days (±3 Days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 39
Participants
  7 days (±3 Days): Yes | 2
  7 days (±3 Days): No | 37
  14 days (±3 Days): number analyzed (Participants) | 36
  14 days (±3 Days): Yes | 2
  14 days (±3 Days): No | 34
  21 days (±3 Days): number analyzed (Participants) | 32
  21 days (±3 Days): Yes | 1
  21 days (±3 Days): No | 31
  28 days (±3 Days): number analyzed (Participants) | 30
  28 days (±3 Days): Yes | 1
  28 days (±3 Days): No | 29

15. Secondary Outcome: Healing of Reference Wound
Description: Wound healed (Yes/No) identified at 7 Days (±3 Days), 14 Days (±3 Days), 21 Days (±3 Days) and 28 day (±3 Days) visits.
Time Frame: 7 days (±3 Days), 14 days (±3 Days), 21 days (±3 Days), 28 days (±3 Days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 40
Participants
  7 days (±3 Days): Yes | 0
  7 days (±3 Days): No | 40
  14 days (±3 Days): number analyzed (Participants) | 36
  14 days (±3 Days): Yes | 1
  14 days (±3 Days): No | 35
  21 days (±3 Days): number analyzed (Participants) | 32
  21 days (±3 Days): Yes | 1
  21 days (±3 Days): No | 31
  28 days (±3 Days): number analyzed (Participants) | 30
  28 days (±3 Days): Yes | 1
  28 days (±3 Days): No | 29

16. Secondary Outcome: Average Dressing Wear Time
Description: Average dressing wear time in days following application
Time Frame: Following dressing application, up to 7 days (±3 Days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 40
days | 4.3 (1.7)

17. Secondary Outcome: Overall Level of Pain on Dressing Application
Description: Level of pain was scored on a scale from 0 to 10 with 0 indicating no pain and 10 indicating the worst pain. Participants provided their level of pain upon each dressing application at each scheduled study visit (7 days, 14 days, 21 days) or at any routine dressing change visit occurring between the scheduled visits.
Time Frame: Immediately after dressing application
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dressings
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 39
Number analyzed (dressings) | 252
score on a scale | 1.1 (2.0)

18. Secondary Outcome: Overall Level of Pain During Treatment
Description: Level of pain was scored on a scale from 0 to 10 with 0 indicating no pain and 10 indicating the worst pain. Participants provided their level of pain during treatment after each dressing application at each scheduled study visit (7 days [ ±3 days], 14 days [ ±3 days], 21 days [ ±3 days]) or at any routine dressing change visit occurring between the scheduled visits.
Time Frame: During treatment (following each dressing application prior to removal), up to 7 days (±3 Days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dressings
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 39
Number analyzed (dressings) | 245
score on a scale | 1.9 (2.6)

19. Secondary Outcome: Overall Level Pain on Dressing Removal
Description: Level of pain was scored on a scale from 0 to 10 with 0 indicating no pain and 10 indicating the worst pain. Participants provided their level of pain on dressing removal for each dressing applied at each scheduled study visit (7 days [ ±3 days], 14 days [ ±3 days], 21 days [ ±3 days]) or at any routine dressing change visit occurring between the scheduled visits.
Time Frame: Immediately upon dressing removal
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dressings
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 39
Number analyzed (dressings) | 246
score on a scale | 1.1 (2.1)

20. Secondary Outcome: Cardiff Wound Impact Schedule (CWIS): Quality of Life at Baseline, 7 Days (±3 Days), 14 Days (±3 Days), 21 Days (±3 Days) and 28 Days (±3 Days)
Description: The Cardiff Wound Impact Schedule (CWIS) was collected at baseline and all study visits. Participants scored on a scale of 0 to 10 their perceived quality of life and satisfaction with quality of life. Higher scores indicate a better outcome.
Time Frame: Baseline, 7 days (±3 Days), 14 days (±3 Days), 21 days (±3 Days), and 28 days (±3 Days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 40
score on a scale
  Quality of Life: Baseline | 6.2 (2.2)
  Quality of Life: 7 days (±3 Days): number analyzed (Participants) | 39
  Quality of Life: 7 days (±3 Days) | 6.3 (2.4)
  Quality of Life: 14 days (±3 Days): number analyzed (Participants) | 39
  Quality of Life: 14 days (±3 Days) | 5.9 (2.4)
  Quality of Life: 21 days (±3 Days): number analyzed (Participants) | 39
  Quality of Life: 21 days (±3 Days) | 6.5 (2.3)
  Quality of Life: 28 days (±3 Days): number analyzed (Participants) | 39
  Quality of Life: 28 days (±3 Days) | 6.6 (2.2)
  Satisfaction with Quality of Life: Baseline: number analyzed (Participants) | 39
  Satisfaction with Quality of Life: Baseline | 6.2 (2.7)
  Satisfaction with Quality of Life: 7 days (±3 Days): number analyzed (Participants) | 39
  Satisfaction with Quality of Life: 7 days (±3 Days) | 6.0 (3.0)
  Satisfaction with Quality of Life: 14 days (±3 Days): number analyzed (Participants) | 39
  Satisfaction with Quality of Life: 14 days (±3 Days) | 6.1 (2.6)
  Satisfaction with Quality of Life: 21 days (±3 Days): number analyzed (Participants) | 39
  Satisfaction with Quality of Life: 21 days (±3 Days) | 6.4 (2.6)
  Satisfaction with Quality of Life: 28 days (±3 Days): number analyzed (Participants) | 39
  Satisfaction with Quality of Life: 28 days (±3 Days) | 6.2 (2.6)

21. Secondary Outcome: Cardiff Wound Impact Schedule (CWIS): Wellbeing, Physical Symptoms & Daily Living, and Social Life at Baseline, 7 (±3 Days), 14 (±3 Days), 21 (±3 Days), and 28 Days (±3 Days)
Description: The Cardiff Wound Impact Schedule (CWIS) was collected at baseline and all study visits. Scores were on a scale from 0 to 100 with a higher score indicating a better outcome across three domains that included:
  * Wellbeing
  * Physical Symptoms & Daily Living
  * Social Life
Time Frame: Baseline, 7 days (±3 Days), 14 days (±3 Days), 21 days (±3 Days), 28 days (±3 Days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 40
score on a scale
  Wellbeing: Baseline | 52.6 (22.4)
  Wellbeing: 7 days (±3 Days): number analyzed (Participants) | 39
  Wellbeing: 7 days (±3 Days) | 55.5 (23.1)
  Wellbeing: 14 days (±3 Days): number analyzed (Participants) | 39
  Wellbeing: 14 days (±3 Days) | 60.8 (23.2)
  Wellbeing: 21 days (±3 Days): number analyzed (Participants) | 39
  Wellbeing: 21 days (±3 Days) | 63.8 (21.0)
  Wellbeing: 28 days (±3 Days): number analyzed (Participants) | 39
  Wellbeing: 28 days (±3 Days) | 61.4 (39)
  Physical Symptoms & Daily Living: Baseline | 69.9 (21.0)
  Physical Symptoms & Daily Living: 7 days (±3 Days): number analyzed (Participants) | 39
  Physical Symptoms & Daily Living: 7 days (±3 Days) | 76.4 (17.0)
  Physical Symptoms & Daily Living: 14 days (±3 Days): number analyzed (Participants) | 39
  Physical Symptoms & Daily Living: 14 days (±3 Days) | 79.2 (17.7)
  Physical Symptoms & Daily Living: 21 days (±3 Days): number analyzed (Participants) | 39
  Physical Symptoms & Daily Living: 21 days (±3 Days) | 81.2 (16.9)
  Physical Symptoms & Daily Living: 28 days (±3 Days): number analyzed (Participants) | 39
  Physical Symptoms & Daily Living: 28 days (±3 Days) | 81.2 (17.4)
  Social Life: Baseline | 72.4 (20.8)
  Social Life: 7 days (±3 Days): number analyzed (Participants) | 39
  Social Life: 7 days (±3 Days) | 77.1 (17.9)
  Social Life: 14 days (±3 Days): number analyzed (Participants) | 39
  Social Life: 14 days (±3 Days) | 82.4 (21.1)
  Social Life: 21 days (±3 Days): number analyzed (Participants) | 39
  Social Life: 21 days (±3 Days) | 86.8 (13.1)
  Social Life: 28 days (±3 Days): number analyzed (Participants) | 39
  Social Life: 28 days (±3 Days) | 85.3 (13.5)

22. Secondary Outcome: Dressing Adherence (Retention)
Description: The investigator determined retention by dressing adherence to the wound at 7 Days (±3 Days), 14 Days (±3 Days), 21 Days (±3 Days) and 28 Day (±3 Days) visits. Dressing adherence reported as the number of participants for each response to the question "Dressing still fully adhered?" from one of the following options:
  * Yes
  * Yes, but with the aid of tape or other material
  * No, study dressing partially adhered
  * No, study dressing not adhered
Time Frame: 7 days (±3 Days), 14 days (±3 Days), 21 days (±3 Days), 28 days (±3 Days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 38
Participants
  7 days (±3 Days): Yes | 20
  7 days (±3 Days): Yes, but with the aid of tape or other material | 12
  7 days (±3 Days): No, study dressing partially adhered | 4
  7 days (±3 Days): No, study dressing not adhered | 2
  14 days (±3 Days): number analyzed (Participants) | 36
  14 days (±3 Days): Yes | 20
  14 days (±3 Days): Yes, but with the aid of tape or other material | 14
  14 days (±3 Days): No, study dressing partially adhered | 1
  14 days (±3 Days): No, study dressing not adhered | 1
  21 days (±3 Days): number analyzed (Participants) | 32
  21 days (±3 Days): Yes | 20
  21 days (±3 Days): Yes, but with the aid of tape or other material | 8
  21 days (±3 Days): No, study dressing partially adhered | 3
  21 days (±3 Days): No, study dressing not adhered | 1
  28 days (±3 Days): number analyzed (Participants) | 29
  28 days (±3 Days): Yes | 21
  28 days (±3 Days): Yes, but with the aid of tape or other material | 5
  28 days (±3 Days): No, study dressing partially adhered | 1
  28 days (±3 Days): No, study dressing not adhered | 2

23. Secondary Outcome: Bunching Up of Dressing
Description: The investigator determined any "bunching up" (i.e., bunching/overlap) of the dressing on the wound at 7 (±3 Days), 14 (±3 Days), 21 (±3 Days) and 28 day visits (±3 Days). Bunching of the dressing reported as the number of participants for each response to "Whether there is any bunching/overlap of dressing" from one of the following options:
  * None
  * Very Little
  * Moderate
  * Excessive
Time Frame: 7 days (±3 Days), 14 days (±3 Days), 21 days (±3 Days), 28 days (±3 Days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 36
Participants
  7 days (±3 Days): None | 29
  7 days (±3 Days): Very Little | 5
  7 days (±3 Days): Moderate | 2
  7 days (±3 Days): Excessive | 0
  14 days (±3 Days): None | 33
  14 days (±3 Days): Very Little | 2
  14 days (±3 Days): Moderate | 0
  14 days (±3 Days): Excessive | 1
  21 days (±3 Days): number analyzed (Participants) | 29
  21 days (±3 Days): None | 21
  21 days (±3 Days): Very Little | 5
  21 days (±3 Days): Moderate | 1
  21 days (±3 Days): Excessive | 2
  28 days (±3 Days): number analyzed (Participants) | 27
  28 days (±3 Days): None | 25
  28 days (±3 Days): Very Little | 1
  28 days (±3 Days): Moderate | 1
  28 days (±3 Days): Excessive | 0

24. Secondary Outcome: Overall Percent of Dressing Lift
Description: Overall percentage of dressing lift for each dressing application was determined from investigator responses following dressing removal at scheduled or routine dressing change visits to the question "Is the study dressing still fully adhered?" The following imputations were used when :
  * If the Investigator answered "Yes" then percentage lift was 0%
  * If the Investigator answered "Study dressing not adhered" then the percentage lift was 100%
  * If "Partially adhered" was selected, then the percentage lift was the percentage indicated in data
Time Frame: Dressing application to removal, up to 7 days (±3 Days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of dressing lift
Units Other Than Participants: dressings
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 38
Number analyzed (dressings) | 250
percentage of dressing lift | 5.8 (20.6)

25. Secondary Outcome: Dressing Comfort During Wear
Description: Dressing comfort at 7 days (±3 Days) , 14 days (±3 Days), 21 days (±3 Days) and 28 day (±3 Days) visits determined by the number of participants with responses to "Dressing comfortable to wear since last visit" from one of the following options:
  * Very comfortable
  * Comfortable
  * Neither comfortable nor uncomfortable
  * Uncomfortable
  * Very uncomfortable
Time Frame: 7 days (±3 Days), 14 days (±3 Days), 21 days( ±3 Days), 28 days (±3 Days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 38
Participants
  7 days (±3 Days): Very comfortable | 20
  7 days (±3 Days): Comfortable | 15
  7 days (±3 Days): Neither comfortable nor uncomfortable | 1
  7 days (±3 Days): Uncomfortable | 1
  7 days (±3 Days): Very uncomfortable | 1
  14 days (±3 Days): number analyzed (Participants) | 35
  14 days (±3 Days): Very comfortable | 19
  14 days (±3 Days): Comfortable | 15
  14 days (±3 Days): Neither comfortable nor uncomfortable | 0
  14 days (±3 Days): Uncomfortable | 1
  14 days (±3 Days): Very uncomfortable | 0
  21 days (±3 Days): number analyzed (Participants) | 31
  21 days (±3 Days): Very comfortable | 16
  21 days (±3 Days): Comfortable | 13
  21 days (±3 Days): Neither comfortable nor uncomfortable | 1
  21 days (±3 Days): Uncomfortable | 1
  21 days (±3 Days): Very uncomfortable | 0
  28 days (±3 Days): number analyzed (Participants) | 30
  28 days (±3 Days): Very comfortable | 17
  28 days (±3 Days): Comfortable | 12
  28 days (±3 Days): Neither comfortable nor uncomfortable | 1
  28 days (±3 Days): Uncomfortable | 0
  28 days (±3 Days): Very uncomfortable | 0

26. Secondary Outcome: Patient Assessment Scale: Leakage
Description: Patient assessment scale completed from baseline visit through end of treatment visits, up to 28 Day (±3 days), using the participant response for each criteria to provide an overall score. Scores ranged from 0 to 10 with 0 indicating a worse outcome and 10 indicating the best outcome. Leakage was determined based on the response to "How have you found your experience in terms of leakage?" where 0 indicated unacceptable level of leakage and 10 indicated no leakage.
Time Frame: Baseline through end of treatment, up to 28 days (±3 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dressings
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 39
Number analyzed (dressings) | 244
score on a scale | 8.6 (2.7)

27. Secondary Outcome: Patient Assessment Scale: Moisture
Description: Patient assessment scale completed from baseline visit through end of treatment visits, up to 28 Day (±3 days), using the participant response for each criteria to provide an overall score. Scores ranged from 0 to 10 with 0 indicating a worse outcome and 10 indicating the best outcome. Moisture was determined based on the response to "How have you found your experience in terms of the feeling of moisture on your skin underneath the dressing" where 0 indicated unacceptable feeling of moisture and 10 indicated no feeling of moisture on the skin.
Time Frame: Baseline through end of treatment, up to 28 days (±3 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dressings
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 39
Number analyzed (dressings) | 244
score on a scale | 8.5 (2.8)

28. Secondary Outcome: Patient Assessment Scale: Odour
Description: Patient assessment scale completed from baseline visit through end of treatment visits, up to 28 Day (±3 days), using the participant response for each criteria to provide an overall score. Scores ranged from 0 to 10 with 0 indicating a worse outcome and 10 indicating the best outcome. Odour was determined based on the response to "How have you found your experience in terms of odour?" where 0 indicated unacceptable level of odour and 10 indicated no odour.
Time Frame: Baseline through end of treatment, up to 28 days (±3 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dressings
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 39
Number analyzed (dressings) | 244
score on a scale | 8.8 (2.5)

29. Secondary Outcome: Patient Assessment Scale: Exudate
Description: Patient assessment scale completed from baseline visit through end of treatment visits, up to 28 Day (±3 days), using the participant response for each criteria to provide an overall score. Scores ranged from 0 to 10 with 0 indicating a worse outcome and 10 indicating the best outcome. Exudate was determined based on the response to "How have you found your experience in terms of visible exudate?" where 0 indicated unacceptable level of visible exudate and 10 indicated no visible exudate.
Time Frame: Baseline through end of treatment, up to 28 days (±3 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dressings
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 39
Number analyzed (dressings) | 243
score on a scale | 6.5 (3.0)

30. Secondary Outcome: Patient Assessment Scale: Protection
Description: Patient assessment scale completed from baseline visit through end of treatment visits, up to 28 Day (±3 days), using the participant response for each criteria to provide an overall score. Scores ranged from 0 to 10 with 0 indicating a worse outcome and 10 indicating the best outcome. Protection was determined based on the response to "How protected did the dressing make your wound feel?" where 0 indicated unacceptable level of protection and 10 indicated very protected.
Time Frame: Baseline through end of treatment, up to 28 days (±3 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dressings
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 39
Number analyzed (dressings) | 244
score on a scale | 8.7 (2.0)

31. Secondary Outcome: Patient Assessment Scale: Comfort
Description: Patient assessment scale completed from baseline visit through end of treatment visits, up to 28 Day (±3 days), using the participant response for each criteria to provide an overall score. Scores ranged from 0 to 10 with 0 indicating a worse outcome and 10 indicating the best outcome. Comfort was determined based on the response to "How have you found your experience in terms of dressing comfort?" where 0 indicated unacceptable level of comfort and 10 indicated very comfortable.
Time Frame: Baseline through end of treatment, up to 28 days (±3 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dressings
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 244
Number analyzed (dressings) | 39
score on a scale | 8.9 (1.7)

32. Secondary Outcome: Patient Assessment Scale: Showering
Description: Patient assessment scale completed from baseline visit through end of treatment visits, up to 28 Day (±3 days), using the participant response for each criteria to provide an overall score. Scores ranged from 0 to 10 with 0 indicating a worse outcome and 10 indicating the best outcome. Comfort was determined based on the response to "How have you found your experience in terms of being able to maintain a normal showering routine? (NA if patient does not have a normal showering routine)" where 0 indicated unacceptable level of impact (unable to bathe) and 10 indicated no negative impact.
Time Frame: Baseline through end of treatment, up to 28 days (±3 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: dressings
Arm/Group | ALLEVYN Gentle Border
Number analyzed (Participants) | 36
Number analyzed (dressings) | 214
score on a scale | 7.8 (3.0)

ADVERSE EVENTS:
Time Frame: Following dressing application to study completion, up to 28 days.
Description: Adverse events were collected for all participants enrolled in the study that received at least one study treatment (i.e., an application of ALLEVYN Gentle Border dressing).
Arm/Group | ALLEVYN Gentle Border
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 4/40
Other Adverse Events (participants affected / at risk) | 10/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALLEVYN Gentle Border (N=40)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) — Possibly related to device
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Subject discontinued from study due to SAE
Urinary tract infection (Infections and infestations) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALLEVYN Gentle Border (N=40)
Wound infection (Infections and infestations) | 3 (3) — Possibly related to study device
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) — Definitely related to study device
Wound complication (Injury, poisoning and procedural complications) | 1 (1) — Subject discontinued due to AE
Skin maceration (Skin and subcutaneous tissue disorders) | 1 (1) — Definitely related to study device
Medical device site erosion (General disorders) | 1 (1) — Definitely related to study device
Urinary retention (Renal and urinary disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
The original study protocol did not specify that participants should have a minimum wound area in the inclusion criteria. As such, several patients were enrolled with particularly small wound areas, limiting the ability to demonstrate suitable wound area reduction. Furthermore, there were eleven participants included who had low levels of exudate at baseline, which was a limiting factor in being able to demonstrate exudate management of the dressing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT03877484/Prot_SAP_000.pdf